CLINICAL TRIAL: NCT07027488
Title: An Open-Label, Phase 1 Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of AB821 in Adult Participants With Locally Advanced or Metastatic Melanoma and Other Solid Tumors
Brief Title: AB821 in Adult Participants With Locally Advanced or Metastatic Solid Tumors
Acronym: Asher-BioAB821
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Asher Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000038990
Record Dates: First submitted 2025-05-19; First posted 2025-06-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Melanoma and Normal or Impaired; Advanced Melanoma
Keywords: AB821; immune-responsive solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AB821 (Experimental): AB821 is intended to be administered as a 30-minute IV infusion every 2 weeks. Dosage is calculated per body weight.
  Interventions: Drug: AB821

INTERVENTIONS:
Drug: AB821 — AB821 will be administered via IV infusion using weight-based dosing. Patients will receive the drug at a dose escalation every two weeks for up to 52 cycles.

SUMMARY:
This study is a first-in-human, open-label, nonrandomized, single center Phase 1 dose-escalation study to assess the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary antitumor activity of AB821 monotherapy given every 2 weeks (Q2W) in participants with recurrent locally advanced or metastatic melanoma and other immune-responsive solid tumors. Immune-responsive solid tumors are defined as those for which immune checkpoint inhibitors form part of the standard-of-care therapy.

DETAILED DESCRIPTION:
This study is a first-in-human, open-label, nonrandomized, single center Phase 1 dose-escalation study to assess the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary antitumor activity of AB821 monotherapy given every 2 weeks (Q2W) in participants with recurrent locally advanced or metastatic melanoma and other immune-responsive solid tumors. Immune-responsive solid tumors are defined as those for which immune checkpoint inhibitors form part of the standard-of-care therapy.

Phase 1 Dose-Escalation: Participants with recurrent locally advanced or metastatic melanoma and immune-responsive solid tumors will be enrolled into dose-escalation cohorts. Patients with melanoma are required to have previously been treated with an inhibitor of PD1/L1, while patients with other solid tumors are required to have had previous systemic treatment regimen that may or may not include an inhibitor of PD1/L1 (n ≥3 for DL3 and above, n=1 for DL1 and 2), to receive AB821 monotherapy to determine MTD or MAD and to select the recommended Phase 1b or Phase 2 dose (RP1bD or RP2D). Participants in dose-escalation cohorts will be enrolled at least 48 hours apart and followed for dose-limiting toxicities for 28 days (completion of two 14-day cycles of treatment).

Dose-Escalation Backfill Cohorts: Based on emerging safety, PK, and pharmacodynamic data, additional participants may be enrolled in backfill cohorts, backfill slots may be used for other tumor types, not only melanoma, upon discussion with the sponsor-investigator at or below dose levels that cleared the dose-limiting toxicity (DLT) assessment and were determined to be safe and tolerable by the Data and Safety Monitoring Board (DSMB). Up to a maximum of 20 total participants may be enrolled in backfill cohorts, at the RP2D or at lower levels deemed efficacious to better assess safety and efficacy based on emerging data. Dose levels and justification are described in Section 4.3.

This study consists of a Screening phase, a Treatment phase, an end of treatment (EOT) Visit, a 30-, 60-, 90- day Safety Follow-up (SFU) phase, and a long-term follow-up (LTFU) phase. Upon completion of the SFU phase post EOT, ongoing safety, disease progression, survival status, and subsequent anticancer therapies will be assessed in the LTFU period.

During the treatment phase, participants who demonstrate disease progression per RECIST criteria may be allowed to continue AB821 if, in the opinion of the treating investigator, the participant is tolerating study treatment and deriving clinical benefit from continuing study treatment. If further progression is noted on subsequent imaging, participants may be allowed to continue on study based on discussion with the sponsor-investigator.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years at the time consent is signed.
2. Ability to provide written informed consent for the study.
3. ECOG PS of 0 or 1.
4. Participants of childbearing potential must not be pregnant at enrollment and agree to comply with contraception requirements. Participants with partners of childbearing potential must also comply with contraception requirements.
5. Adequate organ function as defined below. Specimens must be collected within seven days prior to the start of the study treatment (i.e., Cycle 1 Day 1 [C1D1])
6. Life expectancy of ≥12 weeks, per treating investigator's judgment.
7. For Melanoma participants: Participants with unresectable or metastatic melanoma that have progressed on or after PD 1/PD L1 checkpoint blockade (alone or with either CTLA 4 or LAG 3 checkpoint blockade).

   Note: Participants known to be BRAF V600 mutation-positive; prior therapy with BRAF±MEK inhibitor is at the treating investigator's discretion.
8. For other tumor types: Must have a recurrent histologically or cytologically proven metastatic or locally advanced solid tumor, meeting each of the following:

   1. Tumor that is not amenable to curative treatment with surgery or radiation.
   2. Tumor for which immune checkpoint inhibitors form part of standard-of-care therapy.
   3. Participant has received at least one prior line of systemic anticancer therapy in the recurrent or metastatic setting.
9. Has measurable disease per RECIST v1.1 as assessed by the local site investigator/radiology.

Exclusion Criteria:

1. Has a diagnosis of immunodeficiency.
2. Prior stem cell, bone marrow, or organ transplant.
3. Known history of HIV infection. No HIV testing is required unless mandated by local health authority.
4. History of HBV (defined as HBV surface antigen reactive) or active HCV.
5. Active autoimmune disease (non-immunotherapy induced conditions) that has required systemic treatment in the past two years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic immune-suppressive treatment and is allowed.
6. Active Grade ≥2 diarrhea or enterocolitis.
7. Known active CNS metastases and/or carcinomatous meningitis. Individuals with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression for at least two weeks by repeat imaging, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment).
8. Any other current or previous malignancy within the previous three years except neoplasms that, in the opinion of the treating investigator and with the agreement of the sponsor-investigator, will not interfere with study-specific endpoints, e.g. basal cell carcinoma, localized tumors that have been fully excised with curative intent and no evidence of recurrence or metastasis, prostate cancer that is asymptomatic and does not require therapy other than anti-androgen therapy.
9. Participant is a regular user, as determined by treating investigator judgment (including recreational use), of any illicit drugs or has a recent history (within the last year) of substance abuse (including alcohol), at the time of signing the Informed Consent Form (ICF).
10. Has clinically significant heart disease that affects normal activities, including, unstable angina, or history of congestive heart failure (New York Heart Association Class II IV).
11. History of acute myocardial infarction within the last six months.
12. Has a history of new or worsening thrombosis (DVT/PE, other thrombo-embolic disease) within the last six months.
13. Has a mean QTcF value of >470 ms.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the individuals' participation for the full duration of the study, such that it is not in the best interest of the individual to participate, in the opinion of the treating investigator.
15. Has an active infection, requiring systemic therapy.
16. Has had a severe hypersensitivity reaction to any components of the study treatment or any of their excipients.
17. Is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within seven days prior the first dose of study treatment.
18. Has received more than five prior lines of systemic treatment in the recurrent/metastatic setting.
19. Has received prior radiotherapy within two weeks of start of study treatment or has had a history of radiation pneumonitis.
20. Has a history of grade 3-4 autoimmune myocarditis or a history of Guillain Barre Syndrome.
21. History of congestive heart failure with an ejection fraction < 40%.
22. Participant with NSCLC only: Has received radiation therapy to the lung that is >30 Gy within six months of the first dose of study treatment.
23. Has received previous IL-21 based therapy or prior therapy with AB248
24. Prior systemic anticancer therapy including investigational agents within 4 weeks (or, if shorter, within five half-lives for kinase inhibitors) prior to first dose of study treatment.
25. Major surgery from which the participant has not fully recovered
26. Has received a live or live attenuated vaccine within 30 days
27. Current use of any prohibited concomitant medications.
28. A participant of childbearing potential who has a positive serum pregnancy test within 14 days prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of Dose-Limiting Toxicities (DLTs) in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The primary objective of this outcome measure is to assess the number of participants experiencing dose-limiting toxicities (DLTs) during the study period. DLTs are specific adverse events (AEs) that are considered significant enough to prevent an increase in dose or continuation of treatment.
Frequency of Serious Adverse Events (SAEs) in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This outcome measure aims to record the number of participants who experience serious adverse events (SAEs) while receiving AB821. An SAE is defined as any event that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Frequency of Treatment-Emergent Adverse Events (TEAEs) in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This measure will track the number of participants experiencing treatment-emergent adverse events (TEAEs) during the study. TEAEs are adverse events that emerge following the start of treatment with AB821 and are not present prior to treatment or represent an exacerbation of a pre-existing condition.
Frequency of Adverse Events of Special Interest (AESIs) in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This outcome measure focuses on the number of participants who experience adverse events of special interest (AESIs). AESIs are pre-specified medical occurrences that have been identified as important to monitor due to their potential impact on the risk-benefit profile of AB821.
Frequency of Adverse Events (AEs) Leading to Dose Interruption in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The objective of this measure is to document the number of participants who experience adverse events that result in a temporary interruption of AB821 administration. The interruptions could be due to the severity of the adverse event making it necessary to halt the dosing temporarily.
Frequency of Adverse Events (AEs) Leading to Treatment Discontinuation in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This outcome measure will track the number of participants who experience adverse events leading to the permanent discontinuation of treatment with AB821. These events warrant stopping the treatment altogether to ensure participant safety.
Frequency of Deaths in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The primary objective of this measure is to record the number of participants who die during the study period, irrespective of the cause. This encompasses any deaths occurring within the timeframe of the study and helps to monitor the overall impact of the study treatment on participant mortality.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of AB821 in Serum | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The objective of this outcome measure is to determine the maximum concentration (Cmax) of AB821 in the serum of participants. Cmax represents the highest concentration that AB821 reaches in the bloodstream after administration. This parameter provides important insights into the peak level of drug exposure.
Assessing the immunogenicity of AB821 in patients with advanced melanoma | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The secondary outcome measure will evaluate the immunogenicity of AB821 by monitoring the frequency and titer of anti-drug antibody (ADA) formation against AB821. Additionally, this measure will assess the potential effect of ADA formation on observed safety, pharmacokinetics (PK), and pharmacodynamics (PD) of AB821. The immunogenicity analysis aims to understand the immune response triggered by AB821 and its impact on the therapeutic's overall safety and efficacy profile.
Objective Response Rate (ORR) of AB821 in Patients with Advanced Melanoma | Screening, day 1 of cycle 4 (each cycle is 14 days), end of treatment and at long term follow up
  The objective response rate (ORR) will be determined according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR is defined as the percentage of subjects achieving either a complete response (CR) or partial response (PR).
Duration of Response (DOR) of AB821 in Patients with Advanced Melanoma | Screening, day 1 of cycle 4 (each cycle is 14 days), end of treatment and at long term follow up
  The duration of response (DOR) will be evaluated in subjects who have achieved a complete response (CR) or partial response (PR) as per RECIST v1.1 criteria. DOR is defined as the time from the initial response to documented disease progression or death.
Disease Control Rate (DCR) of AB821 in Patients with Advanced Melanoma | Screening, day 1 of cycle 4 (each cycle is 14 days), end of treatment and at long term follow up
  Disease control rate (DCR) will be assessed according to the RECIST v1.1 criteria. DCR includes the percentage of subjects achieving complete response (CR), partial response (PR), or stable disease (SD).
Progression-Free Survival (PFS) of AB821 in Patients with Advanced Melanoma | Screening, day 1 of cycle 4 (each cycle is 14 days), end of treatment and at long term follow up
  Progression-free survival (PFS) will be measured as the time from the start of treatment with AB821 to the first documentation of disease progression or death from any cause, based on RECIST v1.1 criteria.
Overall Survival (OS) of AB821 in Patients with Advanced Melanoma | Screening, day 1 of cycle 4 (each cycle is 14 days), end of treatment and at long term follow up
  : Overall survival (OS) will be assessed as the time from the start of treatment with AB821 to the time of death from any cause.
Time to Maximum Concentration (tmax) of AB821 in Serum | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This outcome measure aims to identify the time to reach the maximum concentration (tmax) of AB821 in the serum. tmax is the duration it takes after administration for AB821 to reach its peak concentration in the bloodstream. This parameter helps in understanding the absorption rate of the drug.
Area Under the Curve from Time Zero to Last Measurable Concentration (AUC0-last) of AB821 in Serum | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The objective of this measure is to calculate the area under the concentration-time curve from time zero to the last measurable concentration (AUC0-last) of AB821 in serum. AUC0-last provides an integrated measure of the overall exposure to AB821 over time.
Clearance (CL) of AB821 in Serum | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  This outcome measure focuses on determining the clearance (CL) of AB821 from the serum. CL represents the volume of serum from which AB821 is completely removed per unit time. This parameter is crucial for understanding how efficiently the drug is eliminated from the body.
Half-life (t½) of AB821 in Serum | From the date of enrolment to the final follow up visit, approximately two years after the first dose
  The objective of this measure is to determine the half-life (t½) of AB821 in serum. t½ is the time taken for the concentration of AB821 in the serum to reduce to half its maximum level. This parameter gives an indication of the duration AB821 remains active in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No